CLINICAL TRIAL: NCT01781767
Title: Changes in Metabolic Status in Patients With Total Thyroidectomy
Acronym: Thyroid cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-NV-376-CTIL
Record Dates: First submitted 2013-01-27; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Thyroid Cancer
Keywords: UCP2; Thyroid function; Thyroid carcinoma
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood for UCP2 mRNA
Oversight: Data Monitoring Committee: No

SUMMARY:
This study objective is to evaluate the change in mitochondrial uncoupling protein 2 (UCP2) mRNA expression as function of thyroid activity (TSH, T3 and Free T4).

DETAILED DESCRIPTION:
Blood will be drown before thyroidectomy, 2 weeks after the operation and 3-4 month after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with thyroid carcinoma and are going to have total thyroidectomy.
* Patients with unbalanced thyroid hormones.
* Aged 18-65 years at the time of screening.
* Provision of written informed consent.

Exclusion Criteria:

* Patients with Diabetes.
* Patients with any other chronic inflammatory diseases.
* Steroid treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with thyroid carcinoma and are going throgh total thyroidectomy and recive a thyroid replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Changes in UCP2 mRNA concentrations. | Base line (before opporation), 2 weeks after opporation and for after opporation.
  The difference between the result at two weeks and four months compare to base line.

SECONDARY OUTCOMES:
Weight | Approximately 4 months
Resting energy expenditure | Approximatly 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Yen PM. Physiological and molecular basis of thyroid hormone action. Physiol Rev. 2001 Jul;81(3):1097-142. doi: 10.1152/physrev.2001.81.3.1097. PMID 11427693
- [Background] Schwartz HL, Oppenheimer JH. Physiologic and biochemical actions of thyroid hormone. Pharmacol Ther B. 1978;3(3):349-76. doi: 10.1016/s0306-039x(78)80002-6. No abstract available. PMID 203955
- [Background] Brand MD, Esteves TC. Physiological functions of the mitochondrial uncoupling proteins UCP2 and UCP3. Cell Metab. 2005 Aug;2(2):85-93. doi: 10.1016/j.cmet.2005.06.002. PMID 16098826
- [Background] Nicholls DG, Locke RM. Thermogenic mechanisms in brown fat. Physiol Rev. 1984 Jan;64(1):1-64. doi: 10.1152/physrev.1984.64.1.1. No abstract available. PMID 6320232
- [Background] Gjedde S, Gormsen LC, Riis AL, Jorgensen JO, Rungby J, Moller N, Weeke J, Pedersen SB. Reduced expression of uncoupling protein 2 in adipose tissue in patients with hypothyroidism. J Clin Endocrinol Metab. 2010 Jul;95(7):3537-41. doi: 10.1210/jc.2009-0907. Epub 2010 Apr 28. PMID 20427509